CLINICAL TRIAL: NCT02184637
Title: A Five-cohort, Randomized, Open-label, Parallel-group Study to Evaluate the Pharmacokinetics of a Single Dose of Tafenoquine (SB252263) 300mg When Co-administered With the Artemisinin-based Combination Therapies (ACT) Artemether + Lumefantrine (AL) and Dihydroartemisinin + Piperaquine Tetraphosphate (DHA+PQP)
Brief Title: A Study to Evaluate the Pharmacokinetics of a Single Dose of Tafenoquine Co-administered With Either Artemether + Lumefantrine or Dihydroartemisinin + Piperaquine Tetraphosphate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200951
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Malaria, Vivax
Keywords: Malaria; Artemisinin-based Combination Therapies (ACT)
MeSH Terms: conditions — Malaria, Vivax; Malaria | interventions — tafenoquine; artenimol; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1- TQ w/DHA+PQP (Experimental): Tafenoquine (TQ) will be co-administered with Dihydroartemisinin + Piperaquine tetraphosphate (DHA+PQP) on Day 1. DHA+PQP alone will be administered at 24 hours (h) (Day 2) and 48 h (Day 3) post first dose administration.
  Interventions: Drug: Tafenoquine; Drug: Dihydroartemisinin + Piperaquine tetraphosphate
- Cohort 2 - TQ w/AL (Experimental): Tafenoquine co-administered with Artemether + Lumefantrine (AL) on Day 1. AL alone will be administered at 8h (Day 1), 24h and 36h (Day 2), 48h and 60 h (Day 3) post first dose administration.
  Interventions: Drug: Tafenoquine; Drug: Artemether + Lumefantrine
- Cohort 3 - DHA+PQP alone (Experimental): Dihydroartemisinin + Piperaquine tetraphosphate (DHA+PQP) will be administered on Day 1 and at 24 hours (Day 2) and 48 hours (Day 3) post first dose administration
  Interventions: Drug: Dihydroartemisinin + Piperaquine tetraphosphate
- Cohort 4 - AL alone (Experimental): Artemether + Lumefantrine will be administered on Day 1 and 8h, 24 and 36h (Day 2), 48h and 60 h(Day 3) post first dose administration
  Interventions: Drug: Artemether + Lumefantrine
- Cohort 5 - TQ alone (Experimental): A single dose of Tafenoquine will be administered on Day 1
  Interventions: Drug: Tafenoquine

INTERVENTIONS:
Drug: Tafenoquine — A dark pink, capsule-shaped, film-coated tablet containing 150mg tafenoquine. To be administered orally
  Arms: Cohort 1- TQ w/DHA+PQP; Cohort 2 - TQ w/AL; Cohort 5 - TQ alone
Drug: Dihydroartemisinin + Piperaquine tetraphosphate — White, oblong, biconvex, film-coated tablet with a break-line and marked on one side with two "σ" letters containing 320 mg piperaquine tetraphosphate (as the tetrahydrate; PQP) and 40 mg dihydroartemisinin (DHA). To be administered orally
  Arms: Cohort 1- TQ w/DHA+PQP; Cohort 3 - DHA+PQP alone
Drug: Artemether + Lumefantrine — Light yellow, round tablet with "NC" debossed on one side and "CG" on the other, containing 20 mg artemether and 120 mg lumefantrine. To be administered orally
  Arms: Cohort 2 - TQ w/AL; Cohort 4 - AL alone

SUMMARY:
This will be a single-centre, 5-cohort, randomized open-label, parallel-group study in healthy volunteer subjects. This study aims to provide sufficient pharmacokinetic (PK) evidence to support the safe usage of Tafenoquine (TQ) in studies and markets where the Artemisinin-based Combination Therapies (ACTs) are the standard of care for patients with Plasmodium vivax malaria (i.e., co administration with TQ). The objective of this study is to assess the pharmacokinetics, safety and tolerability of TQ when co-administered with the chosen ACTs (AL and DHA + PQP), administered concomitantly in healthy subjects. Specifically, the study will evaluate whether there are drug-drug interactions between TQ and each of the ACTs and if these interactions are considered to be clinically significant. The co-primary objectives of this study are to characterize both the effects of a 300 milligram (mg) single dose of TQ on the pharmacokinetics; changes in (area under the concentration-time curve from 0 to time t) AUC (0-t), AUC (0-infinity), and maximum observed concentration (Cmax) of each of the two Artemisinin-based Combination Therapies (ACT) according to their prescribed dose when co-administered as well as the effects of the ACTs on the PK of TQ.

A total of 120 subjects (24 subjects in each of 5 cohorts) are planned to be enrolled in order to ensure a target sample size of at least 22 subjects completing the study per cohort. All subjects will arrive in the unit at least 24 hours prior to dosing and be discharged after 72-hour post first dose assessments have been completed. Subjects will return for outpatient visits on Days 7, 14, 21, 28, and 56 after first dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s), which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator and GlaxoSmithKline (GSK) Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects whose laboratory values are outside the normal ranges will be excluded from enrolment.
* Male or female aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Alanine Aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5x Upper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* QTcF <440 milliseconds (msec) based on averaged corrected QT interval (QTc) values of triplicate electrocardiogram (ECGs) obtained over a brief recording period at screening and no history of additional risk factors for Torsades des Pointes (e.g., heart failure or family history of Long QT Syndrome).
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-international units per (MIU)/ millilitre (mL) and estradiol <40 picograms (pg)/mL (<147 picomoles (pmol)/liter [L]) is confirmatory]. [Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods, if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.]; Child-bearing potential with negative pregnancy test as determined by serum or urine human chorionic gonadotropin (hCG) test at screening or prior to dosing AND Agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 56-days post first dose. OR has only same-sex partners, when this is her preferred and usual lifestyle.
* Body Mass Index (BMI) within the range 18.5 to 31.0 kilogram/square meter (kg/m^2) (inclusive) and body weight between >=36kilogram (kg) and <=100kg.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject's average triplicate (at screening after approximately 5 minutes at rest in the semi-supine position) systolic blood pressure is outside the range of 80-140 millimeters of mercury (mmHg), or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 40-100 beats per minute (bpm).
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* Lactating females.

Criteria Based Upon Medical Histories:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of thalassaemia; or current or past history of methemoglobinemia or methemoglobin percentage above the reference range at screening.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Consumption of Seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, or grapefruit hybrids from 7 days prior to the first dose of study medication.
* Use of prescription (except female contraception) or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.

Criteria Based Upon Diagnostic Assessments:

* Subjects with a haemoglobin values outside the lower limit of normal range. A single repeat is allowed for eligibility determination.
* Documented phenotypic Glucose-6-phosphate dehydrogenase (G6PD) deficiency, determined by a quantitative assay of enzyme activity. Defined as <70% of locally defined median.
* Potassium <4.0 millimoles (mmol)/L and Magnesium <1.8 mg/ deciliter (dL). Subjects with potassium (K) and magnesium (Mg) values below these screening or on Day-1 may be treated with oral supplementation and be retested for eligibility prior to dosing.
* Cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 30 days prior to screening.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-07-31 (Actual); Primary Completion 2015-04-08 (Actual); Study Completion 2015-04-08 (Actual)

PRIMARY OUTCOMES:
Ratios of Geometric mean (90% [confidence interval] CI) for DHA+PQP AUC and Cmax for treatment groups: Cohort 1 (TQ + DHA+PQP) versus (vs.) cohort 3 (DHA+PQP) | Up to Day 56
  Blood samples will be collected on Day 1 (Pre-dose, 1, 2, 4, 6, 12 hours), Day 2 (24 hours), Day 3 (48, 48.5, 49, 49.5, 50, 51, 52, 54, 56, 60 hours), Day 4 (72 hours), Days 7, 14, 21, 28 and 56.
Ratios of geometric mean [90% CI] for A/DHA/L AUC and Cmax for treatment groups: Cohort 2 (TQ + AL) vs. cohort 4 (AL). | Up to Day 56
  Blood samples will be collected on Day 1 (Pre-dose, 1, 2, 4, 6, 12 hours), Day 2 (24 hours), Day 3 (48, 60, 60.5, 61, 61.5, 62, 64 hours), Day 4 (66, 68, 72 hours), Days 7, 14, 21, 28 and 56.
Ratios of geometric mean [90% CI] for TQ AUC and Cmax for treatment groups: Cohort 1 (TQ + DHA+PQP) vs. cohort 5 (TQ). | Up to Day 56
  Blood samples will be collected on Day 1 (Pre-dose, 1, 2, 4, 6, 12 hours), Day 2 (24 hours), Day 3 (48, 48.5, 49, 49.5, 50, 51, 52, 54, 56, 60 hours), Day 4 (72 hours), Days 7, 14, 21, 28 and 56.
Ratios of geometric mean [90% CI] for TQ AUC and Cmax for treatment groups: Cohort 2 (TQ + AL) vs. cohort 5 (TQ). | Up to Day 56
  Blood samples will be collected on Day 1 (Pre-dose, 1, 2, 4, 6, 12 hours), Day 2 (24 hours), Day 3 (48, 60, 60.5, 61, 61.5, 62, 64 hours), Day 4 (66, 68, 72 hours), Days 7, 14, 21, 28 and 56.

SECONDARY OUTCOMES:
Pharmacokinetic endpoints including changes in time to Cmax (Tmax) and apparent terminal phase half-life (t½) for TQ, as data permit. | Up to Day 56
Pharmacokinetic endpoints including changes in Tmax and t½ for each of the ACTs, as data permit. | Up to Day 56
Changes in safety laboratory measures (including haemoglobin change from baseline [mean of pre-dose and Day-1 results]) | Day -1 to Day 28
  Laboratory assessments will include haematology, clinical chemistry and urinalysis.
Frequency of adverse events (AEs) | Day -1 to Day 56
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Maximum change from baseline in QT interval corrected for heart rate by Fridericia's formula (QTcF) for all cohorts | Day 1 to Day 56
  The baseline measurement will be the average of the triplicate measurements taken on pre-dose Day 1.
Change from baseline in QTcF at 52-hours post-first dose for subjects who receive DHA+PQP (cohort 1 and 3) | Pre-dose (Day 1) and 52-hours post-dose ( Day 3)
  The baseline measurement will be the average of the triplicate measurements taken on pre-dose Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Green JA, Mohamed K, Goyal N, Bouhired S, Hussaini A, Jones SW, Koh GC, Kostov I, Taylor M, Wolstenholm A, Duparc S. Pharmacokinetic Interactions between Tafenoquine and Dihydroartemisinin-Piperaquine or Artemether-Lumefantrine in Healthy Adult Subjects. Antimicrob Agents Chemother. 2016 Nov 21;60(12):7321-7332. doi: 10.1128/AAC.01588-16. Print 2016 Dec. PMID 27697758
- See also: Results for study 200951 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200951?search=study&search_terms=200951#rs
- Available data/document: Dataset Specification: 200951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register